CLINICAL TRIAL: NCT03664349
Title: Improving Communication With Formal/Informal Caregivers Among Older Adults With Dual Sensory Impairment: Feasibility of Hearing Intervention in a Low Vision Rehabilitation Clinic Pilot
Brief Title: Dual Sensory Impairment Low Vision Rehabilitation (LVR) Initiative
Acronym: LVR
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00183648; LVR-F-1 (Other: Other)
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Dual Sensory Impairment of Vision and Hearing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Older Adult Participants and Informal/Formal Caregiver Pairs: A sub-cohort of approximately 10 participant-caregiver pairs will utilize SE9000 and communication strategies over a 4-6-week period between LVR visits.
  Interventions: Device: SuperEar9000
- Older Adult Participants: The pilot cohort of approximately 100 adults over age 60, with vision impairment, will complete the Hearing Handicap Inventory for the Elderly (HHIE), an assessment of perceived impact of hearing impairment, and an objective hearing evaluation.
- Formal/Informal Caregivers: Identified persons who assist willing and eligible older adult pilot participants with two or more ADLs/IADLs.

INTERVENTIONS:
Device: SuperEar9000 — Handheld hearing amplifier, not FDA regulated.
  Groups: Older Adult Participants and Informal/Formal Caregiver Pairs

SUMMARY:
The aims of the Improving Communication with Formal/Informal Caregivers among Older Adults with Dual Sensory Impairment: Feasibility of Hearing Intervention in a Low Vision Rehabilitation Clinic (LVR) are:

Primary aims Aim 1 To characterize prevalence of objective hearing impairment (i.e. DSI) among a clinical LVR population) in older adults (≥60 years) with English proficiency free from moderate to severe depression or cognitive decline using the Hearing Handicap Inventory for the Elderly (HHIE) assessment and an objective hearing evaluation.

Aim 2 To describe the perceived burden of care on primary caregiver (identified people who assist with two or more activities of daily living. instrumental activities of daily living (ADLs/Instrumental activities of daily living (IADLs))of individuals with dual sensory impairment (DSI) among a clinical LVR population in older adults (≥60 years) with English proficiency free from moderate to severe depression or cognitive decline using the Zarit Burden Interview questionnaire and qualitative interview data analyses.

Aim 3 To determine feasibility and benefit of a pilot manualized over-the-counter hearing intervention program on LVR patients to address communication among a DSI population using the Zarit Burden Interview questionnaire.

3A: Describe feasibility based on completion of pilot, drop-out rate, and semi-structured interviews 3B: Describe perceived communication improvements based on semi-structured interviews

DETAILED DESCRIPTION:
The pilot is a prospective cohort study. Approximately 100 participants and their identified people who assist with two or more ADLs/IADLs will be assessed for DSI prevalence and DSI impact on communication. A sub-cohort of 10 participants with DSI will be provided a hearing intervention and followed for 4-6 weeks to assess the over-the-counter hearing intervention program's impact on communication among a DSI population and its identified people who assist with two or more ADLs/IADLs.

Recruitment will be based at the Wilmer Eye Institute (East Baltimore location) LVR clinic. Recruitment efforts will focus on older adults (≥60 years) with English proficiency attending the LVR clinic. Caregivers will be identified based on self-report assistance with at least two ADLs and/or IADLs.

The hearing intervention, for the sub-cohort of 10 individuals with DSI and their identified people who assist with two or more ADLs/IADLs, consists of instruction and best-practices provided by an occupational therapist on the utilization of a handheld amplifier (SuperEar SE9000). Prior to the LVR session with the handheld amplifier, individuals with DSI will complete a daily functioning (ADLs/IADLs) questionnaire (a measure of LVR success). The occupational therapist will give participant a handheld amplifier (SuperEar SE9000) and provide instruction on device use and best-practices (i.e. reducing background noise) to improve communication for the patient-caregiver pairs.

Participant-caregiver pairs will utilize the device and communication strategies over a 4-6-week period between LVR visits. Upon return, pairs will complete semi-structured interviews to elicit information about utilization (successes, barriers), impact on communication, and open qualitative feedback. Participants and caregivers will complete post-intervention functioning questionnaire and Zarit Burden Interview, respectively.

ELIGIBILITY:
Inclusion Criteria- Older Adult Participants

To be eligible for aims 1 & 2 of the study, older adult participants must meet all of the following criteria:

* Age over 60 years. Individuals aged over 60 years at the time of recruitment are eligible for participation.
* Low Vision Rehab Patient/Attendee
* Fluent English Speaker
* Caregiver who reports aiding in 2 or More ADLs/IADLs.
* Residency. Participants must plan to reside in the local area for the pilot duration
* Willingness to participate and adhere to the protocol. Participants must be willing and able to consent to participate in the study, be willing to adhere to the pilot protocol for the duration of the pilot (1 session for aim 1 and aim 2, 2 sessions 4-6 weeks apart for aim 3).

To be eligible for aim 3 of the study, older adult participants must meet the following additional criteria:

* Dual Sensory Impairment (only for aims 2 and 3)
* Hearing Impairment. Participant hearing will be measured by pure tone audiometry a four-frequency test in both ears. Hearing impairment score >=25dB in better ear.

Caregiver (Identified People who Assist with Two or More ADLs/IADLs) Participants

To be eligible for aims 2 & 3 of the study, caregiver participants must meet the following criteria:

• Assist an eligible and willing older adult pilot participant with two or more ADLs/IADLs.

Exclusion Criteria:

Potential candidates for enrollment who meet one or more of the following criteria are excluded from participation in the study:

* Medical contraindication to use handheld amplifier. Because hearing amplifier will be the primary device used in the hearing intervention, participants with medical contraindications to hearing amplifier use are excluded. Contraindication will be determined by pilot audiologist. These may include:
* Active ear infection
* Atresia
* Profound hearing loss beyond the limits of the device
* Asymmetrical hearing loss
* Central hearing loss (i.e. neurologic in origin)
* Free from Vision Impairment. Participants will be excluded who have no vision impairment after refraction on acuity, visual field status and contrast sensitivity as assessed by a low vision rehabilitation clinician.
* Depression. Screened with Center for Epidemiological Studies-Depression (CES-D) score ≥16.
* No participants are excluded based on race or sex.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aim 1 and Aim 2: 100 participants (convenience sample) and their identified people who assist with two or more ADLs/IADLs recruited from Wilmer Eye Institute's LVR clinic Aim 3: sub-cohort of 10 participants with dual sensory impairment and their identified people who assist with two or more ADLs/IADLs
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Dual Sensory Impairment | 1 day
  Measured by the Hearing Handicap Inventory for the Elderly (HHIE), an assessment of perceived impact of hearing impairment, and an objective hearing evaluation (by pure tone audiometry a four-frequency test in both ears. Hearing impairment score >25dB in better ear).
  Total HHIE score: summation of 10 items (0, 2 or 4 points per item, total score range 0 to 40).
  0-8 = no handicap; 10-24 = mild to moderate handicap; 26-40 = severe handicap.

SECONDARY OUTCOMES:
Impact of Dual Sensory Impairment on Formal/informal Caregivers by 12 Question Zarit Burden Interview Questionnaire (Range 0-48, 0-10 mild burden, 10-20 mild to moderate burden, >20 high burden) | 1 day
  Caregivers defined as identified people who assist with two or more ADLs/IADLs). Impact measured by a 12 item Zarit Burden Interview Questionnaire(ZBI-12) to assess burden of care. Total ZBI-12 score: summation of 12 items (0 to 4 points per item, total score range 0 to 48).
  * 0-10: no to mild burden
  * 10-20: mild to moderate burden
  * >20: high burden
Feasibility of Handheld Amplifier on Communication with Formal/Informal Caregivers as assessed by Semi Structured Interviews | 4-6 Weeks
  Feasibility will be measured by semi-structured dyad interviews conducted with formal/informal caregiver and older adult participant pairs. Feasibility will then be determined qualitatively based on participants' response to the interview questions.
Impact of Handheld Amplifier on Caregiver Burden with Formal/Informal Caregivers as assessed by Zarit Burden Interview Questionnaire | 4-6 Weeks
  Impact of hearing amplifier on dyad caregiver burden will be measured with ZBI-12. Total ZBI-12 score: summation of 12 items (0 to 4 points per item, total score range 0 to 48).
  * 0-10: no to mild burden
  * 10-20: mild to moderate burden
  * >20: high burden

CONTACTS AND LOCATIONS:
Overall Officials: Nick Reed, AuD, Principal Investigator — Johns Hopkins Bloomberg School of Medicine
Locations (1):
- Low Vision Rehabilitation Clinic, Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No